CLINICAL TRIAL: NCT00613561
Title: Early Diagnosis and Stem Cell Transplantation for Severe Immunodeficiency Diseases
Acronym: SIDS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Morris Kletzel, MD, Children's Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT 0707; IRB # 2007-13271
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Severe Immunodeficiency Diseases
Keywords: Patients with the Severe Immunodeficiency diseases; Severe Immunodeficiency diseases
MeSH Terms: interventions — fludarabine; Busulfan; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fludarabine, Busulfan, and Anti-Thymocyte Globulin — Patients on this study will receive 5 days of Fludarabine, 1 day of Busulfan Test Dose, 2 Days of Busulfan Regimen Dose, and 4 days of Anti-Thymocyte Globulin
  Other Names: Anti-Thymocyte Globulin is also refered to as ATG.

SUMMARY:
The hypothesis of this study is that children with severe primary immunodeficiencies will benefit from early stem cell transplantation utilizing a reduced intensity conditioning regimen. This regimen is associated with a low risk of complications and will lead to correction of the underlying immunological defects.

ELIGIBILITY:
Inclusion Criteria:

* Must show one of the following diseases:

  * SCIDS
  * Hyper-IgM
  * Wiskott-Aldrich Syndrome
  * Chediak-Higashi and Griscelli Syndromes
  * X-Linked Lymphoproliferative Diseases
  * IPEX Syndrome
  * NEMO Syndrome
  * other severe immunodeficiency diseases not stated above at the discretion of the Principal Investigator
* Informed Consent
* Adequate Renal Function
* Adequate Liver Function
* Adequate Cardiac Function
* Adequate Pulmonary Function
* Adequate Performance Statue
* Adequate Venous Access

Exclusion Criteria:

* Patient/Family has not signed informed consent
* Patient does not have a clear diagnosis of a severe immunodeficiency disease
* A suitable donor for the patient cannot be found
* Patient is HIV positive
* Patient has active Hepatitis B
* Patient is pregnant
* Patient is considered unsuitable for transplant at the discretion of the Principal Investigators or the medical director

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of an optimized reduced intensity conditioning regimen using Fludarabine, Busulfan, and Anti-Thymocyte Globulin in preparing severe immunodeficiency patients for allogeneic hematopoietic progenitor cell transplantation | 5 years

SECONDARY OUTCOMES:
To prospectively follow the natural course of severe immunodeficiency diseases after transplantation | 5 years
To measure the outcomes after stem cell transplantation using the reduced intensity transplant regimen. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Morris Kletzel, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States